CLINICAL TRIAL: NCT03494556
Title: Translating Evidence-Based Chest Pain Decision Aids to the Prehospital Environment
Brief Title: Prehospital Translation of Chest Pain Tools
Acronym: RESCUE
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Cape Fear Valley Mobile Integrated Healthcare Cumberland County EMS (Unknown); New Hanover Regional Medical Center EMS (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00048904
Record Dates: First submitted 2018-04-03; First posted 2018-04-11 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2019-10

CONDITIONS: Acute Coronary Syndrome; Pulmonary Embolism
MeSH Terms: conditions — Acute Coronary Syndrome; Pulmonary Embolism | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No Intervention: Paramedic will use data collected during routine care to complete four risk stratification tools.
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — Paramedic will use data collected during routine care to complete four risk stratification tools.

SUMMARY:
Decision aids such as the HEART Pathway, Emergency Department Assessment of Chest Pain Score (EDACS), Revised Geneva Score and PERC Score have similar ability to accurately risk stratify Emergency Department (ED) patients with possible Acute Coronary Syndrome (ACS) and Pulmonary Embolism (PE) and have become standard practice in the ED setting. This study seeks to determine whether prehospital use of these decision aids is feasible and determine which are the most sensitive and specific for prediction of ACS and PE, respectively.

DETAILED DESCRIPTION:
To accomplish our Specific Aims the study team proposes a prospective, observational pilot study of four rapid risk stratification tools, the HEART Pathway Score, EDACS score, revised Geneva score, and PERC score, among 250 chest pain patients within two large EMS systems. The proposed pilot study has broad-based support from local and state EMS agencies, including Cumberland and New Hanover County EMS agencies. Each tool will be pilot tested and compared in the prehospital setting for feasibility and accuracy. Paramedics will be trained in risk stratification tool use and then will prospectively collect the clinical data needed to calculate each risk stratification score when caring for adults with chest pain. Completed paramedic risk assessments will be used to determine feasibility. Patients will be followed for 30 days to determine occurrence of ACS and PE events and the sensitivity of each risk stratification decision aid will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 21
* Acute non-traumatic chest pain
* Transported by Cumberland or New Hanover County EMS to a local Emergency Department

Exclusion Criteria:

* Patients with evidence of ST elevation myocardial infarction (STEMI) on ECG
* Inter-facility transports (transfers)
* Patients with unstable vital signs
* Prisoners
* Non-english speakers

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being transported to the Emergency Department by Cumberland or New Hanover County EMS.
Sampling Method: Non-Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Determine whether prehospital chest pain decision aid use is feasible. | 24 hours
  Paramedics and blinded Emergency Department providers will be complete four risk stratification tools on a convenience sample of patients with acute chest pain. Inter-rater reliability (kappa) will be determined for each tool.

SECONDARY OUTCOMES:
Compare decision aids to determine which are the most sensitive and specific | 30 days
  Destination hospitals have well established linkages between the prehospital and hospital Electronic Medical Record (EMR) facilitating patient outcome ascertainment. Data will be abstracted from the EMR to determine occurrence of 30 day study outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Stopyra, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Cape Fear Valley Mobile Integrated Healthcare Cumberland County EMS, Fayetteville, North Carolina
  - New Hanover Regional Medical Center EMS, Wilmington, North Carolina

IPD SHARING:
Plan to Share IPD: No
At this time, the study does not have plans to share individual participant data, including data dictionaries, with other researchers.

REFERENCES:
- [Background] Owens PL, Barrett ML, Gibson TB, Andrews RM, Weinick RM, Mutter RL. Emergency department care in the United States: a profile of national data sources. Ann Emerg Med. 2010 Aug;56(2):150-65. doi: 10.1016/j.annemergmed.2009.11.022. Epub 2010 Jan 15. PMID 20074834
- [Background] Lowthian JA, Cameron PA, Stoelwinder JU, Curtis A, Currell A, Cooke MW, McNeil JJ. Increasing utilisation of emergency ambulances. Aust Health Rev. 2011 Feb;35(1):63-9. doi: 10.1071/AH09866. PMID 21367333
- [Background] Pittet V, Burnand B, Yersin B, Carron PN. Trends of pre-hospital emergency medical services activity over 10 years: a population-based registry analysis. BMC Health Serv Res. 2014 Sep 10;14:380. doi: 10.1186/1472-6963-14-380. PMID 25209450
- [Background] Saddichha S, Saxena MK. Is every chest pain a cardiac event? : an audit of patients with chest pain presenting to emergency services in India. Intern Emerg Med. 2009 Jun;4(3):235-9. doi: 10.1007/s11739-009-0246-3. Epub 2009 Apr 15. PMID 19367468
- [Background] Burman RA, Zakariassen E, Hunskaar S. Acute chest pain - a prospective population based study of contacts to Norwegian emergency medical communication centres. BMC Emerg Med. 2011 Jul 21;11:9. doi: 10.1186/1471-227X-11-9. PMID 21777448
- [Background] Mahler SA, Miller CD, Hollander JE, Nagurney JT, Birkhahn R, Singer AJ, Shapiro NI, Glynn T, Nowak R, Safdar B, Peberdy M, Counselman FL, Chandra A, Kosowsky J, Neuenschwander J, Schrock JW, Plantholt S, Diercks DB, Peacock WF. Identifying patients for early discharge: performance of decision rules among patients with acute chest pain. Int J Cardiol. 2013 Sep 30;168(2):795-802. doi: 10.1016/j.ijcard.2012.10.010. Epub 2012 Oct 30. PMID 23117012
- [Background] Mahler SA, Riley RF, Hiestand BC, Russell GB, Hoekstra JW, Lefebvre CW, Nicks BA, Cline DM, Askew KL, Elliott SB, Herrington DM, Burke GL, Miller CD. The HEART Pathway randomized trial: identifying emergency department patients with acute chest pain for early discharge. Circ Cardiovasc Qual Outcomes. 2015 Mar;8(2):195-203. doi: 10.1161/CIRCOUTCOMES.114.001384. Epub 2015 Mar 3. PMID 25737484
- [Background] Thang ND, Sundstrom BW, Karlsson T, Herlitz J, Karlson BW. ECG signs of acute myocardial ischemia in the prehospital setting of a suspected acute coronary syndrome and its association with outcomes. Am J Emerg Med. 2014 Jun;32(6):601-5. doi: 10.1016/j.ajem.2014.03.006. Epub 2014 Mar 15. PMID 24731933
- [Background] Mahler SA, Hiestand BC, Goff DC Jr, Hoekstra JW, Miller CD. Can the HEART score safely reduce stress testing and cardiac imaging in patients at low risk for major adverse cardiac events? Crit Pathw Cardiol. 2011 Sep;10(3):128-33. doi: 10.1097/HPC.0b013e3182315a85. PMID 21989033
- [Background] Flaws D, Than M, Scheuermeyer FX, Christenson J, Boychuk B, Greenslade JH, Aldous S, Hammett CJ, Parsonage WA, Deely JM, Pickering JW, Cullen L. External validation of the emergency department assessment of chest pain score accelerated diagnostic pathway (EDACS-ADP). Emerg Med J. 2016 Sep;33(9):618-25. doi: 10.1136/emermed-2015-205028. Epub 2016 Jul 12. PMID 27406833
- [Background] Than M, Flaws D, Sanders S, Doust J, Glasziou P, Kline J, Aldous S, Troughton R, Reid C, Parsonage WA, Frampton C, Greenslade JH, Deely JM, Hess E, Sadiq AB, Singleton R, Shopland R, Vercoe L, Woolhouse-Williams M, Ardagh M, Bossuyt P, Bannister L, Cullen L. Development and validation of the Emergency Department Assessment of Chest pain Score and 2 h accelerated diagnostic protocol. Emerg Med Australas. 2014 Feb;26(1):34-44. doi: 10.1111/1742-6723.12164. Epub 2014 Jan 15. PMID 24428678
- [Background] Le Gal G, Righini M, Roy PM, Sanchez O, Aujesky D, Bounameaux H, Perrier A. Prediction of pulmonary embolism in the emergency department: the revised Geneva score. Ann Intern Med. 2006 Feb 7;144(3):165-71. doi: 10.7326/0003-4819-144-3-200602070-00004. PMID 16461960
- [Background] Kline JA, Mitchell AM, Kabrhel C, Richman PB, Courtney DM. Clinical criteria to prevent unnecessary diagnostic testing in emergency department patients with suspected pulmonary embolism. J Thromb Haemost. 2004 Aug;2(8):1247-55. doi: 10.1111/j.1538-7836.2004.00790.x. PMID 15304025
- [Background] Havas S. The ACCORD Trial and control of blood glucose level in type 2 diabetes mellitus: time to challenge conventional wisdom. Arch Intern Med. 2009 Jan 26;169(2):150-4. doi: 10.1001/archinternmed.2008.518. No abstract available. PMID 19171811
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Katus HA, Lindahl B, Morrow DA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S. Third universal definition of myocardial infarction. Circulation. 2012 Oct 16;126(16):2020-35. doi: 10.1161/CIR.0b013e31826e1058. Epub 2012 Aug 24. No abstract available. PMID 22923432
- [Background] Pollack CV, Schreiber D, Goldhaber SZ, Slattery D, Fanikos J, O'Neil BJ, Thompson JR, Hiestand B, Briese BA, Pendleton RC, Miller CD, Kline JA. Clinical characteristics, management, and outcomes of patients diagnosed with acute pulmonary embolism in the emergency department: initial report of EMPEROR (Multicenter Emergency Medicine Pulmonary Embolism in the Real World Registry). J Am Coll Cardiol. 2011 Feb 8;57(6):700-6. doi: 10.1016/j.jacc.2010.05.071. PMID 21292129